CLINICAL TRIAL: NCT06672315
Title: Transesophageal Echocardiography in Pre-hospital Cardiac Arrest Patients; TAPCAP
Brief Title: Application of Transesophageal Echocardiography in Pre-hospital Cardiac Arrest Patients
Acronym: TAPCAP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jen-Tang Sun (Other)
Responsible Party: Sponsor-Investigator, Jen-Tang Sun, Director of Emergency Surgery, Far Eastern Memorial Hospital
Organization: Far Eastern Memorial Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 113027-F
Record Dates: First submitted 2024-09-30; First posted 2024-11-04 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-03

CONDITIONS: Out-of-hospital Cardiac Arrest (OHCA)
Keywords: Left Ventricular Outflow Tract; Transesophageal Echocardiography; TEE; LVOT; OHCA
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest | interventions — Echocardiography, Transesophageal

STUDY DESIGN:
Intervention Model Description: Patients aged 18 years or older who have experienced out-of-hospital cardiac arrest (OHCA) due to non-traumatic causes
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- Performing TEE (Experimental): In this group of patients, transesophageal echocardiography (TEE) will be performed to confirm optimal chest compression positioning while utilizing a mechanical chest compression device.
  Interventions: Diagnostic Test: transesophageal echocardiography
- not performing TEE (No Intervention): In this group of patients, transesophageal echocardiography (TEE) will not be performed, and the mechanical chest compression device will be positioned at the intersection of the nipple line and the sternum.

INTERVENTIONS:
Diagnostic Test: transesophageal echocardiography — Confirmation of chest compression positioning via transesophageal echocardiography (TEE)
  Arms: Performing TEE

SUMMARY:
The Use of Point-of-Care Ultrasound (POCUS), Transthoracic Echocardiography (TTE), and Transesophageal Echocardiography (TEE) in Cardiac Arrest and Acute Coronary Syndrome Patients

Studies have shown that POCUS can rapidly change the management in nearly 80% of cases in emergency settings, particularly in environments such as war zones and disaster relief. TTE is highly sensitive in diagnosing acute coronary syndromes and can effectively rule out myocardial infarction. In cardiac arrest patients, TTE assists in determining cardiac activity and identifying reversible causes, such as pericardial tamponade and pneumothorax. However, TTE can be affected by suboptimal image quality due to factors like chest compression in out-of-hospital cardiac arrest (OHCA) patients.

In Taiwan's emergency medical system, EMT-Ps (paramedics) undergo approximately one year of training, which enables them to provide emergency care, including ultrasound examinations, before hospital arrival. Research on pre-hospital cardiac arrest has shown that most ultrasound applications can be completed within 3 minutes and do not significantly increase on-scene time.

TEE, though advantageous for its high-quality imaging and ability to reduce interruptions during chest compressions, faces challenges in pre-hospital emergency applications due to specialized training and equipment requirements. However, a study in Vienna, Austria, demonstrated that TEE could be performed and yield high-quality images in most pre-hospital cases, with an average examination time of 5.1 minutes.

Several hospitals in Taiwan have begun training personnel in TEE, emphasizing the importance of establishing TEE image registries for large-scale, effective research analysis. However, these efforts also face challenges related to resources and collaboration. The research team has over three years of experience using TEE in the emergency department to examine OHCA patients, and a three-year study will be conducted to validate the efficacy of pre-hospital TEE in cardiac arrest patients.

DETAILED DESCRIPTION:
Background:

The application of Point-of-Care Ultrasound (POCUS), Transthoracic Echocardiography (TTE), and Transesophageal Echocardiography (TEE) in cardiac arrest and acute coronary syndrome has evolved with technological advancements. POCUS, in particular, has been recognized for its ability to change clinical management in nearly 80% of emergency cases, such as war and disaster scenarios. TTE is highly sensitive in diagnosing acute coronary syndromes and can effectively rule out myocardial infarction. It also plays a crucial role in identifying reversible causes in cardiac arrest patients, like pericardial tamponade and pneumothorax, but its image quality can be compromised during chest compressions in out-of-hospital cardiac arrest (OHCA) patients. TEE, on the other hand, offers superior image quality and reduces interruptions during chest compressions but requires specialized training and equipment.

Currently, Taiwan's emergency medical system allows EMT-P personnel, after a year of training, to perform pre-hospital ultrasounds, including POCUS, for OHCA patients. Research has shown that most ultrasound applications can be completed in under 3 minutes without significantly increasing on-scene time. TEE's use in pre-hospital emergencies has also been validated in international studies, such as those from Vienna, which demonstrated TEE's feasibility in providing clear diagnostic images during pre-hospital cardiac arrest care.

Research Methods:

This study aims to assess the feasibility and efficacy of TEE in pre-hospital cardiac arrest care through a randomized controlled trial over three years.

Study Design:

The study will be conducted in two phases:

Phase 1: A prospective observational feasibility study involving 60 patients to assess the practical application of TEE in pre-hospital settings.

Patients aged 18 or older. Non-traumatic OHCA patients.

Exclusion Criteria:

Signs of obvious death. Patients with DNR orders. Patients for whom TEE is contraindicated (e.g., esophageal tumors). Patients requiring ECPR.

Training and Implementation:

Emergency department staff and EMT teams will undergo specialized training, including TEE workshops and simulations. The TEE procedure will be performed after establishing the airway and during mechanical chest compressions using a LUCAS device.

Data Collection:

Data will include patient demographics, emergency response times, CPR parameters, and TEE imaging results. Outcomes such as return of spontaneous circulation (ROSC) and neurological recovery will be tracked.

Randomization:

The RCT phase will utilize cluster randomization based on bi-weekly intervals, ensuring random and balanced patient groupings for intervention and control.

Sample Size Estimation:

Based on prior studies and statistical analysis, each group will require 93 patients to detect significant differences, with a total of 186 patients over the course of 24 months.

Expected Results:

The study anticipates that the use of TEE in pre-hospital cardiac arrest care will:

Provide high-quality cardiac images during CPR. Facilitate accurate identification of reversible causes of cardiac arrest. Improve the overall effectiveness of CPR through real-time feedback. Demonstrate the feasibility of integrating TEE into pre-hospital emergency protocols without significantly delaying patient transport.

The primary outcome is the proportion of cases where TEE ensures optimal chest compression. Secondary outcomes include the rate of sustained ROSC, time to ROSC, and neurological outcomes.

Conclusion:

This study will provide valuable insights into the feasibility and impact of TEE in pre-hospital cardiac arrest management. It will serve as the foundation for future large-scale research and contribute to improving survival rates and neurological outcomes in OHCA patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Patients with out-of-hospital cardiac arrest (OHCA)
3. Non-traumatic cause of cardiac arrest

Exclusion Criteria:

1. Presence of obvious signs of death, such as decapitation, rigor mortis, livor mortis, or decomposition.
2. Family explicitly expresses a Do Not Attempt Resuscitation (DNR) order, or the patient has a documented refusal of resuscitation.
3. Any condition that contraindicates the use of transesophageal echocardiography (TEE), such as esophageal tumors, preventing probe insertion.
4. Patients eligible for ECPR (Extracorporeal Cardiopulmonary Resuscitation) treatment.
5. Spontaneous circulation has already been stabilized before performing TEE.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-12-30 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility of using TEE to assist OHCA patients in pre-hospital emergency treatment | 30 days after cardiac arrest or upon the patient's death, whichever came first
  Feasibility of using TEE to assist OHCA patients in pre-hospital emergency treatment. The proportion of successfully ensuring LV compression during prehospital CPR.

SECONDARY OUTCOMES:
Sustained return of spontaneous circulation (sustained ROSC) lasting approximately 20 minutes | Patient sustained ROSC for 20 minutes after
Time from the start of resuscitation to the first return of spontaneous circulation (ROSC) | 1 minute after patient first ROSC
  Time from the start of resuscitation to the first return of spontaneous circulation (ROSC)
Any ROSC rate | 1 minute after patient ROSC
  Any ROSC rate
Favorable neurologic outcome with discharge to home (Cerebral Performance Category 1 or 2) | Up to 6 months after discharge date
  Record the patient's neurological outcome at the time of discharge
End-tidal carbon dioxide (EtCO2) | One hour after arriving at the hospital
  End-tidal carbon dioxide (EtCO2) values during the resuscitation process.

CONTACTS AND LOCATIONS:
Locations (1):
- Far Eastern Memorinal Hospital and New Taipei City fire department, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
Name and email

REFERENCES:
- [Background] Krammel M, Hamp T, Hafner C, Magnet I, Poppe M, Marhofer P. Feasibility of resuscitative transesophageal echocardiography at out-of-hospital emergency scenes of cardiac arrest. Sci Rep. 2023 Nov 16;13(1):20085. doi: 10.1038/s41598-023-46684-x. PMID 37973909
- [Background] Hermann M, Hafner C, Scharner V, Hribersek M, Maleczek M, Schmid A, Schaden E, Willschke H, Hamp T. Remote real-time supervision of prehospital point-of-care ultrasound: a feasibility study. Scand J Trauma Resusc Emerg Med. 2022 Mar 24;30(1):23. doi: 10.1186/s13049-021-00985-0. PMID 35331304
- [Background] Reed MJ, Gibson L, Dewar A, Short S, Black P, Clegg GR. Introduction of paramedic led Echo in Life Support into the pre-hospital environment: The PUCA study. Resuscitation. 2017 Mar;112:65-69. doi: 10.1016/j.resuscitation.2016.09.003. Epub 2016 Sep 13. PMID 27638418
- [Background] Botker MT, Vang ML, Grofte T, Kirkegaard H, Frederiksen CA, Sloth E. Implementing point-of-care ultrasonography of the heart and lungs in an anesthesia department. Acta Anaesthesiol Scand. 2017 Feb;61(2):156-165. doi: 10.1111/aas.12847. PMID 28066904
- [Background] Clattenburg EJ, Wroe P, Brown S, Gardner K, Losonczy L, Singh A, Nagdev A. Point-of-care ultrasound use in patients with cardiac arrest is associated prolonged cardiopulmonary resuscitation pauses: A prospective cohort study. Resuscitation. 2018 Jan;122:65-68. doi: 10.1016/j.resuscitation.2017.11.056. Epub 2017 Nov 23. PMID 29175356
- [Background] Huis In 't Veld MA, Allison MG, Bostick DS, Fisher KR, Goloubeva OG, Witting MD, Winters ME. Ultrasound use during cardiopulmonary resuscitation is associated with delays in chest compressions. Resuscitation. 2017 Oct;119:95-98. doi: 10.1016/j.resuscitation.2017.07.021. Epub 2017 Jul 25. PMID 28754527
- [Background] El Sayed MJ, Zaghrini E. Prehospital emergency ultrasound: a review of current clinical applications, challenges, and future implications. Emerg Med Int. 2013;2013:531674. doi: 10.1155/2013/531674. Epub 2013 Sep 19. PMID 24171113
- [Background] Chin EJ, Chan CH, Mortazavi R, Anderson CL, Kahn CA, Summers S, Fox JC. A pilot study examining the viability of a Prehospital Assessment with UltraSound for Emergencies (PAUSE) protocol. J Emerg Med. 2013 Jan;44(1):142-9. doi: 10.1016/j.jemermed.2012.02.032. Epub 2012 May 16. PMID 22595631
- [Background] Hussein L, Rehman MA, Jelic T, Berdnikov A, Teran F, Richards S, Askin N, Jarman R; SHoC Investigators and the Resuscitative TEE Collaborative Registry Investigators. Transoesophageal echocardiography in cardiac arrest: A systematic review. Resuscitation. 2021 Nov;168:167-175. doi: 10.1016/j.resuscitation.2021.08.001. Epub 2021 Aug 12. PMID 34390824
- [Background] Breitkreutz R, Price S, Steiger HV, Seeger FH, Ilper H, Ackermann H, Rudolph M, Uddin S, Weigand MA, Muller E, Walcher F; Emergency Ultrasound Working Group of the Johann Wolfgang Goethe-University Hospital, Frankfurt am Main. Focused echocardiographic evaluation in life support and peri-resuscitation of emergency patients: a prospective trial. Resuscitation. 2010 Nov;81(11):1527-33. doi: 10.1016/j.resuscitation.2010.07.013. PMID 20801576
- [Background] Hayhurst C, Lebus C, Atkinson PR, Kendall R, Madan R, Talbot J, Ross P, Lewis D. An evaluation of echo in life support (ELS): is it feasible? What does it add? Emerg Med J. 2011 Feb;28(2):119-21. doi: 10.1136/emj.2009.084202. Epub 2010 Oct 4. PMID 20921017
- [Background] Long B, Alerhand S, Maliel K, Koyfman A. Echocardiography in cardiac arrest: An emergency medicine review. Am J Emerg Med. 2018 Mar;36(3):488-493. doi: 10.1016/j.ajem.2017.12.031. Epub 2017 Dec 16. PMID 29269162
- [Background] Rybicki FJ, Udelson JE, Peacock WF, Goldhaber SZ, Isselbacher EM, Kazerooni E, Kontos MC, Litt H, Woodard PK. 2015 ACR/ACC/AHA/AATS/ACEP/ASNC/NASCI/SAEM/SCCT/SCMR/SCPC/SNMMI/STR/STS Appropriate Utilization of Cardiovascular Imaging in Emergency Department Patients With Chest Pain: A Joint Document of the American College of Radiology Appropriateness Criteria Committee and the American College of Cardiology Appropriate Use Criteria Task Force. J Am Coll Cardiol. 2016 Feb 23;67(7):853-79. doi: 10.1016/j.jacc.2015.09.011. Epub 2016 Jan 22. No abstract available. PMID 26809772
- [Background] Atkinson P, Bowra J, Milne J, Lewis D, Lambert M, Jarman B, Noble VE, Lamprecht H, Harris T, Connolly J; and members of the International Federation of Emergency Medicine Sonography in Hypotension and Cardiac Arrest working group: Romolo Gaspari, MD, PhD; Ross Kessler, MD; Christopher Raio, MD; Paul Sierzenski, MD; Beatrice Hoffmann, MD; Chau Pham, MD; Michael Woo, MD; Paul Olszynski, MD; Ryan Henneberry, MD; Oron Frenkel, MD; Jordan Chenkin, MD; Greg Hall, MD; Louise Rang, MD; Maxime Valois, MD; Chuck Wurster, MD; Mark Tutschka, MD; Rob Arntfield, MD; Jason Fischer, MD; Mark Tessaro, MD; J. Scott Bomann, DO; Adrian Goudie, MB; Gaby Blecher, MB; Andree Salter, MB; Michael Rose, MB; Adam Bystrzycki, MB; Shailesh Dass, MB; Owen Doran, MB; Ruth Large, MB; Hugo Poncia, MB; Alistair Murray, MB; Jan Sadewasser, MD; Raoul Breitkreutz, MD; Hong Chuen Toh, MB; Arif Alper Cevik, MD; Ang Shiang Hu, MB; Larry Melniker, MD, MS. International Federation for Emergency Medicine Consensus Statement: Sonography in hypotension and cardiac arrest (SHoC): An international consensus on the use of point of care ultrasound for undifferentiated hypotension and during cardiac arrest. CJEM. 2017 Nov;19(6):459-470. doi: 10.1017/cem.2016.394. Epub 2016 Dec 21. PMID 27998322
- [Background] Leonardi M, Condous G. A pictorial guide to the ultrasound identification and assessment of uterosacral ligaments in women with potential endometriosis. Australas J Ultrasound Med. 2019 Aug 9;22(3):157-164. doi: 10.1002/ajum.12178. eCollection 2019 Aug. PMID 34760552
- [Background] Stawicki SP, Howard JM, Pryor JP, Bahner DP, Whitmill ML, Dean AJ. Portable ultrasonography in mass casualty incidents: The CAVEAT examination. World J Orthop. 2010 Nov 18;1(1):10-9. doi: 10.5312/wjo.v1.i1.10. PMID 22474622
- [Background] Moore CL, Copel JA. Point-of-care ultrasonography. N Engl J Med. 2011 Feb 24;364(8):749-57. doi: 10.1056/NEJMra0909487. No abstract available. PMID 21345104
- [Background] Atkinson PR, Milne J, Diegelmann L, Lamprecht H, Stander M, Lussier D, Pham C, Henneberry R, Fraser JM, Howlett MK, Mekwan J, Ramrattan B, Middleton J, van Hoving DJ, Peach M, Taylor L, Dahn T, Hurley S, MacSween K, Richardson LR, Stoica G, Hunter S, Olszynski PA, Lewis DA. Does Point-of-Care Ultrasonography Improve Clinical Outcomes in Emergency Department Patients With Undifferentiated Hypotension? An International Randomized Controlled Trial From the SHoC-ED Investigators. Ann Emerg Med. 2018 Oct;72(4):478-489. doi: 10.1016/j.annemergmed.2018.04.002. Epub 2018 Jun 2. PMID 29866583